CLINICAL TRIAL: NCT04130620
Title: Red Blood Cell Validation of Magnesium Deficiency as Determined by a Muscle Stretch Test
Brief Title: Validation of the Magnesium Muscle Stretch Test
Acronym: PAKMGTEST
Status: Completed | Type: Observational
Sponsor: Anthony Rosner (Other)
Collaborators: William Maykel, D.C., Wellness Medicine (Other)
Responsible Party: Sponsor-Investigator, Anthony Rosner, Co-Principal Investigator-Sponsor, William Maykel, D.C., Wellness Medicine
Organization: William Maykel, D.C., Wellness Medicine (Other)
Other Study IDs: 1004401
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Magnesium Deficiency
Keywords: Magnesium deficiency; Applied Kinesiology
MeSH Terms: conditions — Magnesium Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Applied Kinesiology — An Applied Kinesiology muscle test will be supplemented by a single blood draw for validation.
  Other Names: :Blood Draw

SUMMARY:
Professional Applied Kinesiology (PAK) is a system which attempts to evaluate numerous aspects of health (structural, chemical, and mental) by the manual testing of muscles, combined with other standard methods of diagnosis. It leads to a variety of conservative, noninvasive treatments which involves joint manipulations or mobilizations, myofascial therapies, cranial techniques, meridian and acupuncture skills, clinical nutrition and dietary management, counseling skills, evaluating environmental irritants, and various reflex techniques. The expanded validity of the manual muscle test has been extensively described.elsewhere, including by one of the Co-Principal Investigators (Anthony Rosner). Details of Applied Kinesiology and its adjunctive procedures are prescribed by an International College of Applied Kinesiology Board of Examiners, cited for its scholarly and scientific activities.

A convenience sample of 40 patients, ages 18-75, will be administered the magnesium muscle stretch test with blood drawn at the time of the individual's visit. For the muscle test, uniformity of the examiner's force application is to be confirmed with a force transducer, while the clinician's judgment as to whether the muscle test is positive (facilitated) or negative (inhibited) will be confirmed by electrogoniometry, the procedures for both the force transducer and electrogoniometer having been established by one of the Co-PIs (Anthony Rosner) previously. The blood sample is to be submitted to LabCorp for the measurement of red blood cell levels of magnesium. Coded results of the muscle test and magnesium blood levels are to be correlated by an experienced statistician who is blinded to the patient's identity.

DETAILED DESCRIPTION:
A convenience sample of 40 patients, ages 18-75. is to be selected from those attending the services of Dr. William Maykel at his office in Auburn, Massachusetts. Consenting patients are be given an informed consent form approved by a contract institutional review board (PearlIRB), which they are to sign and return indicating that they fully understand the scope and logistics of the proposed research with the right to withdraw at any time without reprisals. Research subjects will undergo the manual muscle stretch test administered by Dr. William Maykel. Specifically, the stretch test is performed as follows:

1. The patient is seated. The right anterior serratus muscle is tested. The doctor asks the patient to hold the right arm straight out at a 90 degree angle with the thumb pointed toward the ceiling.
2. The muscle test is 5/5.
3. The patient is instructed to raise his or her arm straight up to the ceiling, stretching the anterior serratus muscle. The arm is then brought back to the original test position at a 90 degree angle with the thumb up.
4. The muscle is then retested. If it is now 3/5, this represents a positive magnesium stretch test.
5. The procedure is repeated on one or two other muscles to solidify the diagnostic presence of insufficient magnesium.

Immediately afterward, the patient's blood is drawn by a licensed phlebotomist with samples submitted to LabCorp to determine red blood cell magnesium contents (and other trace metals for future investigations).

Results of the muscle test (inhibited or facilitated) are to be paired with the respective blood magnesium levels and shared with each participant. They will be coded to protect the patient's identity identity and submitted to an experienced statistician for correlation, the results either supporting or refuting the hypothesis which stated that the muscle stretch test is a rapid, inexpensive, and readily available screening test for magnesium deficiency. Correlation will be a binary process, based upon (i) normal or deficient levels of magnesium based upon the muscle testing, and (ii) normal blood cell ranges of magnesium established by the reference laboratory. The identity of patients will be known only to the research staff and kept within a locked file in Dr. Maykel's office for 5 years before being discarded. It will not be shared in any presentations or publications of research results.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, speak, and understand English

Exclusion Criteria:

* Disability Cognitive impairments History of bleeding disorder Known arterial aneurysm Current pregnancy Involvement in healthcare litigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Routinely scheduled patients of William Maykel, D.C., receiving chiropractic adjustments, manual muscle testing, and/or nutritional therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Applied Kinesiology muscle test result | Change from baseline muscle position to one after test is concluded (3 seconds)
  Facilitated (strong) or inhibited (weak)
Red blood cell level | Baseline
  Routine blood draw and red blood cell magnesium measurement in mcg/g

CONTACTS AND LOCATIONS:
Overall Officials: Anthony L Rosner, Ph.D., Principal Investigator — Medical Information Services
Locations (1):
- Malchar Chiropractic Wellness Center, Warwick, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD with patient's identity masked according to HIPAA regulations will be tabulated and described in publications and presentations at professional society meetings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD with patient's identity masked according to HIPAA regulations will be shared, starting March 2020 when it will be submitted in manuscript form for publication. It will continue to be shared with resubmissions/and/or professional society meetings for 5 years following that date.
Access Criteria: IPD sharing will occur with patient's identity masked with a statistician, professional journal reviewers and editors, and individuals in professional healthcare who are colleagues and/or who attend professional society meetings.

REFERENCES:
- [Result] Rosner AL, Cuthbert SC. Applied kinesiology: distinctions in its definition and interpretation. J Bodyw Mov Ther. 2012 Oct;16(4):464-87. doi: 10.1016/j.jbmt.2012.04.008. Epub 2012 May 11. PMID 23036878
- [Result] Volpe SL. Magnesium in disease prevention and overall health. Adv Nutr. 2013 May 1;4(3):378S-83S. doi: 10.3945/an.112.003483. PMID 23674807
- [Result] Altura BM, Altura BT. Magnesium and contraction of arterial smooth muscle. Microvasc Res. 1974 Mar;7(2):145-55. doi: 10.1016/0026-2862(74)90001-6. No abstract available. PMID 4363012
- [Result] Potter JD, Robertson SP, Johnson JD. Magnesium and the regulation of muscle contraction. Fed Proc. 1981 Oct;40(12):2653-6. PMID 7286246
- [Result] Bothe G, Coh A, Auinger A. Efficacy and safety of a natural mineral water rich in magnesium and sulphate for bowel function: a double-blind, randomized, placebo-controlled study. Eur J Nutr. 2017 Mar;56(2):491-499. doi: 10.1007/s00394-015-1094-8. Epub 2015 Nov 18. PMID 26582579
- [Result] Mayer ML, Westbrook GL, Guthrie PB. Voltage-dependent block by Mg2+ of NMDA responses in spinal cord neurones. Nature. 1984 May 17-23;309(5965):261-3. doi: 10.1038/309261a0. PMID 6325946
- [Result] Nowak L, Bregestovski P, Ascher P, Herbet A, Prochiantz A. Magnesium gates glutamate-activated channels in mouse central neurones. Nature. 1984 Feb 2-8;307(5950):462-5. doi: 10.1038/307462a0. PMID 6320006
- [Result] Morris ME. Brain and CSF magnesium concentrations during magnesium deficit in animals and humans: neurological symptoms. Magnes Res. 1992 Dec;5(4):303-13. PMID 1296767
- [Result] de Baaij JH, Hoenderop JG, Bindels RJ. Magnesium in man: implications for health and disease. Physiol Rev. 2015 Jan;95(1):1-46. doi: 10.1152/physrev.00012.2014. PMID 25540137
- [Result] Yavuz Y, Mollaoglu H, Yurumez Y, Ucok K, Duran L, Tunay K, Akgun L. Therapeutic effect of magnesium sulphate on carbon monoxide toxicity-mediated brain lipid peroxidation. Eur Rev Med Pharmacol Sci. 2013 Feb;17 Suppl 1:28-33. PMID 23436663
- [Result] Feldman Z, Gurevitch B, Artru AA, Oppenheim A, Shohami E, Reichenthal E, Shapira Y. Effect of magnesium given 1 hour after head trauma on brain edema and neurological outcome. J Neurosurg. 1996 Jul;85(1):131-7. doi: 10.3171/jns.1996.85.1.0131. PMID 8683262
- [Result] Hasturk AE, Harman F, Arca T, Sargon M, Kilinc K, Kaptanoglu E. Neuroprotective effect of magnesium sulfate and dexamethasone on intrauterine ischemia in the fetal rat brain: ultrastructural evaluation. Turk Neurosurg. 2013;23(5):666-71. doi: 10.5137/1019-5149.JTN.8541-13.1. PMID 24101316
- [Result] Solomon D, Bunegin L, Albin M. The effect of magnesium sulfate administration on cerebral and cardiac toxicity of bupivacaine in dogs. Anesthesiology. 1990 Feb;72(2):341-6. doi: 10.1097/00000542-199002000-00021. PMID 2301766
- [Result] Held K, Antonijevic IA, Kunzel H, Uhr M, Wetter TC, Golly IC, Steiger A, Murck H. Oral Mg(2+) supplementation reverses age-related neuroendocrine and sleep EEG changes in humans. Pharmacopsychiatry. 2002 Jul;35(4):135-43. doi: 10.1055/s-2002-33195. PMID 12163983
- [Result] Zieve FJ, Freude KA, Zieve L. Effects of magnesium deficiency on protein and nucleic acid synthesis in vivo. J Nutr. 1977 Dec;107(12):2178-88. doi: 10.1093/jn/107.12.2178. PMID 925766
- [Result] Kenney MA, McCoy H, Williams L. Effects of magnesium deficiency on strength, mass, and composition of rat femur. Calcif Tissue Int. 1994 Jan;54(1):44-9. doi: 10.1007/BF00316289. PMID 8118753
- [Result] Bogoroch R, Belanger LF. Skeletal effects of magnesium deficiency in normal, ovariectomized, and estrogen-treated rats. Anat Rec. 1975 Nov;183(3):437-47. doi: 10.1002/ar.1091830308. PMID 1200332
- [Result] Rude RK, Singer FR, Gruber HE. Skeletal and hormonal effects of magnesium deficiency. J Am Coll Nutr. 2009 Apr;28(2):131-41. doi: 10.1080/07315724.2009.10719764. PMID 19828898
- [Result] Salem M, Kasinski N, Munoz R, Chernow B. Progressive magnesium deficiency increases mortality from endotoxin challenge: protective effects of acute magnesium replacement therapy. Crit Care Med. 1995 Jan;23(1):108-18. doi: 10.1097/00003246-199501000-00019. PMID 8001362
- [Result] Andrieux-Domont C, Le van Hung. Effects of magnesium deficiency on reproduction in the white rat. Br J Nutr. 1973 Mar;29(2):203-10. doi: 10.1079/bjn19730095. No abstract available. PMID 4693557
- [Result] Stokic E, Romani A, Ilincic B, Kupusinac A, Stosic Z, Isenovic ER. Chronic Latent Magnesium Deficiency in Obesity Decreases Positive Effects of Vitamin D on Cardiometabolic Risk Indicators. Curr Vasc Pharmacol. 2018;16(6):610-617. doi: 10.2174/1570161115666170821154841. PMID 28828979
- [Result] Rosanoff A, Weaver CM, Rude RK. Suboptimal magnesium status in the United States: are the health consequences underestimated? Nutr Rev. 2012 Mar;70(3):153-64. doi: 10.1111/j.1753-4887.2011.00465.x. Epub 2012 Feb 15. PMID 22364157
- [Result] Whang R. Magnesium deficiency: pathogenesis, prevalence, and clinical implications. Am J Med. 1987 Mar 20;82(3A):24-9. doi: 10.1016/0002-9343(87)90129-x. PMID 3565424
- [Result] Schmitt WH Jr, Leisman G. Correlation of applied kinesiology muscle testing findings with serum immunoglobulin levels for food allergies. Int J Neurosci. 1998 Dec;96(3-4):237-44. doi: 10.3109/00207459808986471. PMID 10069623
- [Result] Schmitt WH Jr, Yanuck SF. Expanding the neurological examination using functional neurologic assessment: part II neurologic basis of applied kinesiology. Int J Neurosci. 1999 Mar;97(1-2):77-108. doi: 10.3109/00207459908994304. PMID 10681119
- [Result] Leisman G, Shambaugh P, Ferentz AH. Somatosensory evoked potential changes during muscle testing. Int J Neurosci. 1989 Mar;45(1-2):143-51. doi: 10.3109/00207458908986227. PMID 2714940
- [Result] Lawson A, Calderon L. Interexaminer agreement for applied kinesiology manual muscle testing. Percept Mot Skills. 1997 Apr;84(2):539-46. doi: 10.2466/pms.1997.84.2.539. PMID 9106846
- [Result] Cuthbert SC, Goodheart GJ Jr. On the reliability and validity of manual muscle testing: a literature review. Chiropr Osteopat. 2007 Mar 6;15:4. doi: 10.1186/1746-1340-15-4. PMID 17341308
- See also: International College of Applied Kinesiology-USA — http://www.icakusa.com